CLINICAL TRIAL: NCT05213260
Title: Flipped Classroom Approach Application to Clinical Skills for Preclinical Medical Students
Brief Title: Effectiveness of Flipped Classroom in Clinical Skills Teaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dar Al Uloom University (Other)
Responsible Party: Principal Investigator, Dr. Einas Yousef, Principal Investigator, Dar Al Uloom University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro 22030013
Record Dates: First submitted 2022-01-04; First posted 2022-01-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Medical Education; Simulation Based Learning
Keywords: Preclinical medical students; Clinical skills learning; Flipped classroom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Flipped Teaching Method Group) (Experimental): Flipped classroom for intervention group:
  The students allotted to the flipped classroom teaching approach will receive the pre-session learning materials (video access links) three days prior to the clinical case session through their institutional email addresses. Students will be encouraged to complete the assigned tasks before coming to class.
  The session will start by reviewing the objectives, discussing the difficult points they have in the preparation materials, and answering any question. They also will be shortly briefed about how the scenario would run. They will have a fixed time to take the cardiovascular history, perform examination, order appropriate investigations, reach a differential diagnosis, and formulate a treatment plan. During the session, the instructor will evaluate these students at each level of clinical case-solving. Finally, post-session survey will be disseminated via email to know the students' perception of the flipped teaching.
  Interventions: Other: Flipped Teaching method
- Control group (Traditional Method Group) (No Intervention): This group of students, included 20 participants, will be briefed by the instructors for 30 minutes immediately before the clinical skill session about the clinical case which will include: history taking, examination, investigations, diagnosis, and treatment plan. Following that, there will be time for practice and discussion amongst the students on a high-fidelity manikin. Of note, these students will not receive any pre-session teaching material as the intervention group.

INTERVENTIONS:
Other: Flipped Teaching method — Before the clinical skill laboratory session, the students will receive the learning materials that they have to read and assimilate before the in-class part which will include interactive, discussion-oriented, and practice-oriented activities.
  Arms: intervention group (Flipped Teaching Method Group)

SUMMARY:
College of Medicine, DAU University, is a private college, located in Riyadh, Saudi Arabia, which launched its activity in 2013. Since that time, there is a continuous increase in the number of students, especially during the last three years after the graduation of the first batch, which is not associated with the recruitment of new faculty. Of course, this increase in the number of students has affected greatly the interaction between the instructors and the students. Another challenging point is the short time assigned for most of the preclinical years' courses as most of our blocks have 5-8 weeks duration with a lot of work needed to be done to help students demonstrate mastery of the intended learning outcomes. As a response to these problems, the investigators sought to pilot testing flipping the classroom of clinical skill sessions as a new educational approach in our college.

DETAILED DESCRIPTION:
The current study will be conducted in the Clinical skill and simulation center of the College of Medicine, Dar Al Uloom University, Riyadh, Saudi Arabia. Students will be informed that participation was anonymous, voluntary, and this intervention will be an extracurricular activity that will not count to their actual grades.

Participants To reduce performance bias, a group of 40 third-year medical students (academic year 2020-2021) will randomly assigned to flipped or traditional learning sessions. These students had already completed the Cardiovascular block in the second semester of their second year. The cardiovascular block (6 credit hours, 6 weeks) contents handle all the subjects related to cardiovascular system from the view of the basic medical sciences such as anatomy, physiology, biochemistry, microbiology and pathology, and pharmacology. Besides, clinical medical sciences integrated in this block as clinical skill sessions that run synchronously with the lectures and focus on the application of relevant medical practice using clinical skills and simulation center. They took a total of three sessions in the block, each running for 2 hours.

To ensure that each student has an equal chance of getting exposed to any of the teaching approaches used in our study, the students will be randomized into interventional and control groups. The attendance registers of all third-year students will be considered, from which every third student will be selected making a total of 40. Out of these the first 20 formed the intervention group and the second 20 were considered as the control group. To avoid the Hawthorne effect (change of the participants' behavior in response to their awareness of being observed), the students will be blinded to their groups and will be unaware of when and what will be assessed throughout the skill lab sessions [1]. Notably, both control and interventional groups will be supervised by the same medical teachers, have the same scenario, and same simulated patients. They will finally evaluated by the same instructors based on a well-structured checklist.

Preparation of flipped classroom materials Three instructors worked to prepare the study materials, for the application of the flipped classroom teaching methodology in the clinical skill and simulation center for the preclinical students. The learning objectives of the cardiovascular clinical case were identified. We gathered the following relevant, high-quality videos from YouTube: Cardiovascular History Taking Key Symptoms OSCE Guide, Cardiovascular Examination - OSCE Guide, Heart murmur sounds, and Blood pressure measurement - OSCE guide. Moreover, short PowerPoint presentations including teaching materials (investigations and treatment) and pertinent to the clinical case were created and saved as videos. Of note, all included videos are shorter than 10 minutes in duration. All these materials were uploaded into the freely accessible EdPuzzle software to embed our own questions at appropriate places in the videos. The EdPuzzle platform helped to assign these videos to a group of students and get hassle-free analytics: see who watched the video, who didn't understand the lesson and who did a good job. Students can re-watch the video as many times as they need at their own pace, while we can easily check their progress from our account. Reports of student answers will be prepared by teacher prior to face-to-face session, and logs of the students' interaction with the videos will be monitored by the teacher.

ELIGIBILITY:
Inclusion Criteria:

* Third-year medical students
* Successfully completed the cardiovascular block.
* Agreed to participate in the study

Exclusion Criteria:

* Refused to participate in the study
* Did not successfully completed the cardiovascular block.
* All students from the clinical phase and UPP (preparatory phase)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Assessing students' performance | During the session while performing the skills
  Students in the control and study group will be assessed by the tutors based on a certain checklist

SECONDARY OUTCOMES:
Perception of students included in the flipped classroom | immediately after the flipped teaching session
  the students will be requested to fill a questionnaire about their perception with the flipped teaching in skill lab.

CONTACTS AND LOCATIONS:
Overall Officials: Einas M Yousef, Ph.D., Principal Investigator — College of Medicine, Dar Al Uloom University
Locations (1):
- College of Medicine, Dar Al Uloom University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No